CLINICAL TRIAL: NCT07276334
Title: Outpatient vs. Inpatient Surgery for Distal Radius Fractures: A Prospective Randomized Trial
Brief Title: Same Day Discharge Vs. Hospitalization for Operative Fixation of Distal Radius Fractures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Ofir Vinograd, Principal investigator, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASF-25-0106
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Distal Radius Fracture Fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same-day-discharge (Experimental)
  Interventions: Procedure: early release from hospital
- Hospitalized (Active Comparator)
  Interventions: Procedure: Day after surgery release

INTERVENTIONS:
Procedure: early release from hospital — Same day discharge of patients undergoing distal radius operative fixation
  Arms: Same-day-discharge
Procedure: Day after surgery release — release of patients one day after surgery
  Arms: Hospitalized

SUMMARY:
The goal of this clinical trial is to examine the results for same-day discharge after distal radius operative fixation in adult pupolation. The main questions it aims to answer are:

Is same day discharge safe and effective for distal radius fractures? Are the functional and patient reported outcome measures results different between same day discharge and hospitalized patients? Researchers will compare same day discharge patients with jospitalized patients to see if there are any differences between the groups

Participants will:

* undergo surgery
* atend outpatient clinical follow up visits
* answer dedicated questioneres

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and
* diagnosed with a DRF requiring surgical intervention and
* booked for surgery

Exclusion Criteria:

* Refusal to participate in the study
* lack of follow-up
* incomplete clinical or radiologic documentation
* significant cardiac or pulmonary comorbidities
* inadequate social support at home

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire, | from surgery to one year after
  A self-report tool (0-100) measuring upper limb function, where higher scores mean more disability,

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical Center, Ẕerifin, Israel, Israel